CLINICAL TRIAL: NCT03138135
Title: HOME Study: Evaluation of a Combination Support Package to Increase Uptake of Pre-exposure Prophylaxis and HIV/STI Testing Among Young Black and Latino MSM in the San Francisco Bay Area.
Brief Title: HOME Study: a Combination Support Package to Increase Uptake of PrEP and HIV/STI Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Public Health Foundation Enterprises, Inc. (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); San Francisco Department of Public Health (Other Government); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Susan Buchbinder, Director, Bridge HIV, Public Health Foundation Enterprises, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 16-20492; R01AI104309 (NIH)
Record Dates: First submitted 2017-04-14; First posted 2017-05-03 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: HIV Prevention; Sexually Transmitted Diseases; Pre-Exposure Prophylaxis
Keywords: PrEP; HIV prevention; Risk reduction; STI prevention; Home HIV testing; HIV testing; STI testing
MeSH Terms: conditions — Sexually Transmitted Diseases; Risk Reduction Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The Intervention group will receive the HOME Study intervention.
  Interventions: Behavioral: HOME Study intervention
- Control (Active Comparator): The Control group will receive standard of care.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: HOME Study intervention — Access to home HIV test kits, home STI self-collection kits, the HOME Study website, and the SexPro HIV risk assessment tool.
  Arms: Intervention
Behavioral: Control — Counseling about the importance of quarterly HIV/STI testing and a PrEP information pamphlet.
  Arms: Control

SUMMARY:
Home HIV self-testing has been FDA approved and allows users to read their own HIV test results at home, while home sexually transmitted infection (STI) test self-collection allows men to use a swab at home and mail it in for testing. The purpose of this study is to learn how Men who have Sex with Men (MSM) use these new testing options, a set of online support tools, and the option to test with someone to support them (a testing "buddy").

We will also evaluate whether the online tools help these men to connect with HIV prevention services such as Pre-Exposure Prophylaxis (PrEP) if they test HIV negative, and to HIV care services if they test HIV positive.

DETAILED DESCRIPTION:
Participants will be randomized 2:1 after enrollment to the intervention and control condition. Data obtained from this study will be used to inform the further tailoring and distribution of an intervention for young Black and Latino MSM to increase utilization of home HIV self-testing and linkage to HIV treatment and Pre-Exposure Prophylaxis (PrEP).

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as Black or Latino.
* Report anal sex with at least one male sex partner in the prior 12 months.
* HIV negative by self-report.
* Currently own a cell phone.
* Willing and able to provide written informed consent.

Exclusion Criteria:

* Inadequate contact information for follow-up.
* In a mutually monogamous sexual relationship for the past 12 months.
* Currently taking PrEP.
* Does not have reliable access to the Internet.
* Does not live, work, or play in the San Francisco Bay Area.
* Planning to move out of the Bay Area during the 9 month study period.
* Previously participated in the HOME Pilot study.
* Any medical, psychiatric, or social condition, or occupational, or other responsibility that, in the judgment of the investigator, would make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Cisgender male
Enrollment: 104 (Actual)
Dates: Start 2017-01-09 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Efficacy of the HOME package to support linkage to PrEP or HIV care | 9 months
  Between-arm differences in initiation of PrEP; qualitative evaluation of linkage to HIV care.
Efficacy of the HOME package to increase HIV and STI testing frequency. | 9 months
  The proportion of participants reporting HIV and STI testing rates between visits.

SECONDARY OUTCOMES:
Feasibility of the individual components of the study intervention. | 9 months
  Combined analysis of overall use of study intervention: Usage of home HIV self-testing, with and without buddies, as well as STI-self collection; Proportion of participants who log-in to the HOME Study site at least once, distribution of numbers of log-ins, and use of HOME Study pages, as measured by numbers of clicks and views for each page.
Acceptability of the HOME package to support linkage to HIV care or PrEP. | 9 months
  Acceptability scores from online questionnaires and the distribution of repeated scores at follow-up timepoints.

OTHER OUTCOMES:
Who uses home HIV self-testing and home STI self-collection. | 9 months
  Testing and self-collection rates by occasion, age, county, race/ethnicity, and prior testing history. Aggregate descriptive analysis.
Who uses a buddy. | 9 months
  Differences in testing with a buddy by occasion, age, county, race/ethnicity, and prior testing history. Aggregate descriptive analysis.
Use of HIV prevention services. | 9 months
  Proportion of HIV uninfected participants who attend group or individual counseling services.

CONTACTS AND LOCATIONS:
Overall Officials: Hyman Scott, MD, MPH, Principal Investigator — Public Health Foundation Enterprises; San Francisco Department of Public Health; Susan Buchbinder, MD, Principal Investigator — Public Health Foundation Enterprises; San Francisco Department of Public Health
Locations (1):
- Bridge HIV, San Francisco Department of Public Health, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Bridge HIV Health Equity Studies homepage — http://helpfighthiv.org